CLINICAL TRIAL: NCT00755274
Title: Annual Study for Serum Collection and Evaluation of Safety and Immunogenicity Among Healthy Children Receiving Fluzone® Influenza Virus Vaccine (2008-2009 Formulation)
Brief Title: Annual Study for Serum Collection for Immunogenicity and Safety Evaluation in Healthy Children Receiving Fluzone®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC40
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Results first posted 2010-04-01 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza; Orthomyxoviridae Infections
Keywords: Influenza; Orthomyxoviruses; Orthomyxoviridae Infections; Influenza vaccine
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Primed (Experimental): Have received 2 or more lifetime Flu Vaccinations Prior to Visit 1
  Interventions: Biological: Influenza Virus Vaccine No Preservative: Pediatric Dose
- Group 2: Naive/Inadequately Primed (Experimental): Never Received or Received Only 1 Lifetime Flu Vaccination Prior to Visit 1
  Interventions: Biological: Influenza Virus Vaccine No Preservative: Pediatric Dose

INTERVENTIONS:
Biological: Influenza Virus Vaccine No Preservative: Pediatric Dose — 0.25 mL, IM (age 6-35 months) or 0.5 mL, IM (age 36-59 months)
  Other Names: Fluzone®
  Arms: Group 1: Primed
Biological: Influenza Virus Vaccine No Preservative: Pediatric Dose — 0.25 mL, IM (age 6-35 months) or 0.5 mL, IM (age 36-59 months)
  Other Names: Fluzone®
  Arms: Group 2: Naive/Inadequately Primed

SUMMARY:
Primary Objective:

To provide the Center for Biologics Evaluation and Research (CBER) with sera collected from healthy children receiving the 2008-2009 formulation of the inactivated, split-virion influenza vaccine Fluzone® for further study.

Observational Objectives:

To describe the safety of the 2008-2009 pediatric formulation of Fluzone® vaccine, administered in a one- or two-dose schedule in accordance with Advisory Committee on Immunization Practices (ACIP) recommendations, in children ≥ 6 months to < 5 years of age.

To describe the immunogenicity of the 2008-2009 pediatric formulation of Fluzone® vaccine, administered in a one- or two-dose schedule in accordance with ACIP recommendations, in children ≥ 6 months to < 5 years of age.

DETAILED DESCRIPTION:
The Advisory Committee on Immunization Practices (ACIP) has in recent years recommended that all healthy children aged 6 through 59 months receive influenza vaccine. Because of the growing emphasis on influenza immunization of infants and young children, Center for Biologics Evaluation and Research (CBER) has expressed interest in receiving sera from children who have been vaccinated with the current formulation of Fluzone® vaccine. These sera will be tested to evaluate each individual's immune response to the current formulation of Fluzone® vaccine and will also be used to evaluate circulating influenza strains in order to support formulation recommendations for the subsequent year (particularly for influenza B strains, which predominantly affect the young).

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥ 6 months to < 5 years of age.
* Participant is considered to be in good health on the basis of reported medical history and a limited history-directed physical examination.
* Parent/legal acceptable representative is willing and able to bring the subject to the scheduled visits and to comply with the study procedures during the entire duration of the study.
* Parent/legal acceptable representative is willing and able to provide informed consent.
* Subject was born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2.5 kg (5.5 lbs).

Exclusion Criteria:

* Reported allergy to egg proteins, chicken proteins, or any other constituent of the vaccine.
* History of severe adverse event to any influenza vaccine.
* Laboratory-confirmed influenza infection or vaccination against influenza in the 6 months preceding enrollment in the study.
* Any vaccination scheduled between Visit 1 and Visit 2.
* Planned participation in any other interventional clinical trial during participation in the study.
* Known or suspected impairment of immunologic function or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Personal or immediate family history of congenital immune deficiency.
* Developmental delay, neurologic disorder, or seizure disorder.
* Chronic medical, congenital, or developmental disorder.
* Known Human immunodeficiency virus (HIV)-positive mother.
* Prior personal history of Guillain-Barré syndrome.
* Any condition which, in the opinion of the Investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular (IM) vaccination.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi pasteur Inc.
Locations (1):
- Norfolk, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 15 September to 1 October 2008 in 1 clinical center in the US.
Pre-assignment Details: A total of 32 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Primed Group: Participants had received 2 or more lifetime influenza vaccinations prior to Visit 1. They received a single intramuscular dose of Fluzone® (0.25 mL for those aged 6-35 months and 0.5 mL for those aged 36-59 months) at Visit 1.
- Naive/Inadequately Primed Group: Participants never received or received only 1 lifetime influenza vaccination prior to Visit 1. They received one intramuscular dose of Fluzone® (0.25 mL for those aged 6-35 months and 0.5 mL for those aged 36-59 months) at Visit 1 and a second dose at Visit 2.
Period: Overall Study
Arm/Group | Primed Group | Naive/Inadequately Primed Group
Started | 24 | 8
Completed | 24 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primed Group | Naive/Inadequately Primed Group | Total
Number analyzed (Participants) | 24 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 8 | 32
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 32.8 (10.52) | 22.1 (10.36) | 30.1 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 4 | 17
  Male | 11 | 4 | 15
Region of Enrollment [Number; unit: participants]
  United States | 24 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Reactions After Fluzone® Vaccination 1
Description: Solicited local reactions: Tenderness, pain, erythema, and swelling. Systemic reactions: Fever (temperature), vomiting, crying abnormal, drowsiness, appetite lost, irritability, headache, malaise, and myalgia.
Time Frame: Day 0 to Day 3 post-vaccination 1
Population: Safety analysis was on all enrolled and vaccinated participants with available post-vaccination 1 data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Primed Group | Naive/Inadequately Primed Group
Number analyzed (Participants) | 24 | 8
Participants
  Any Solicited Injection Site Reaction | 10 | 2
  Any Tenderness | 2 | 1
  Grade 3 Tenderness (Cries When Limb Is Moved) | 0 | 0
  Any Pain | 8 | 1
  Grade 3 Pain (Incapacitating) | 0 | 0
  Any Erythema | 0 | 2
  Grade 3 Erythema (≥ 5 cm) | 0 | 0
  Any Swelling | 1 | 1
  Grade 3 Swelling (≥ 5 cm) | 0 | 0
  Any Solicited Systemic Reaction | 12 | 4
  Any Fever | 2 | 2
  Grade 3 Fever (> 103.1 ºF) | 0 | 0
  Any Vomiting | 0 | 1
  Grade 3 Vomiting (≥ 6 Episodes per 24 hours) | 0 | 0
  Any Crying Abnormal | 0 | 0
  Grade 3 Crying Abnormal (> 3 hours) | 0 | 0
  Any Drowsiness | 4 | 0
  Grade 3 Drowsiness (Sleeps most of time) | 0 | 0
  Any Appetite Lost | 1 | 0
  Grade 3 Appetite Lost (Refuses ≥ 3 meals/feeds) | 0 | 0
  Any Irritability | 2 | 1
  Grade 3 Irritability (Inconsolable) | 0 | 0
  Any Headache | 1 | 1
  Grade 3 Headache (Prevents daily activities) | 0 | 0
  Any Malaise | 4 | 1
  Grade 3 Malaise (Prevents daily activities) | 0 | 0
  Any Myalgia | 6 | 0
  Grade 3 Myalgia (Prevents daily activities) | 0 | 0

2. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Antibodies to Vaccine Influenza Strains Determined by Hemagglutination Inhibition (HAI) Assay After Fluzone® Vaccination
Time Frame: Day 28 post-single dose or Day 21 post-Dose 2
Population: Geometric mean titers (GMTs) to the Influenza vaccine antibodies were determined in the per-protocol population.
  One each of the enrolled participants in the Primed and Naive groups, respectively, did not have valid post-vaccination serology test data.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Primed Group | Naive/Inadequately Primed Group
Number analyzed (Participants) | 23 | 7
Titers
  H1N1 Flu A/Brisbane/59/2007 IVR-148 Pre, All | 54.8 [28.5 to 105.5] | 8.6 [3.5 to 21.3]
  H3N2 Flu A/Uruguay/716/2007/X175-C Pre, All | 24.5 [12.7 to 47.6] | 10.5 [3.0 to 37.1]
  B Flu B/Florida/04/2006 Pre, All | 5.3 [4.9 to 5.8] | 5.0 [5.0 to 5.0]
  H1N1 Flu A/Brisbane/59/2007 IVR-148 Pre, 6-35 mo | 46.5 [21.5 to 101.0] | 8.6 [3.5 to 21.3]
  H3N2 Flu A/Uruguay/716/2007/X175-C Pre, 6-35 mo | 17.9 [8.4 to 38.3] | 10.5 [3.0 to 37.1]
  B Flu B/Florida/04/2006 Pre, 6-35 mo | 5.2 [4.8 to 5.7] | 5.0 [5.0 to 5.0]
  H1N1 Flu A/Brisbane/59/2007 IVR-148 Post, All | 320.0 [218.7 to 468.3] | 168.1 [70.0 to 403.9]
  H3N2 Flu A/Uruguay/716/2007/X175-C Post, All | 510.5 [305.2 to 854.0] | 226.3 [62.8 to 815.5]
  B Flu B/Florida/04/2006 Post, All | 26.2 [13.1 to 52.4] | 31.2 [14.0 to 69.5]
  H1N1 Flu A/Brisbane/59/2007 IVR-148 Post, 6-35 mo | 320.0 [196.8 to 520.4] | 168.1 [70.0 to 403.9]
  H3N2 Flu A/Uruguay/716/2007/X175-C Post, 6-35 mo | 424.1 [223.5 to 804.7] | 226.3 [62.8 to 815.5]
  B Flu B/Florida/04/2006 Post, 6-35 mo | 18.3 [8.2 to 40.9] | 31.2 [14.0 to 69.5]

3. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Antibodies to Vaccine Influenza Strains Determined by Hemagglutination Inhibition (HAI) Assay After Fluzone® Vaccination
Time Frame: Day 28 post-single dose or Day 21 post-Dose 2
Population: Geometric mean titers (GMTs) to the Influenza vaccine antibodies were determined in the per-protocol population. (Data is part of Outcome 3, no data were generated for the Naive/Inadequately Primed Group).
  One of the enrolled participants in the Primed group did not have valid post-vaccination serology test data.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Primed Group | Naive/Inadequately Primed Group
Number analyzed (Participants) | 23 | 0
Titers
  H1N1 Flu A/Brisbane/59/2007 IVR-148, Pre 36-59 mo | 84.8 [16.0 to 448.2] |
  H3N2 Flu A/Uruguay/716/2007/ X175-C, Pre 36-59 mo | 56.6 [12.3 to 260.2] |
  B Flu B/Florida/04/2006, Pre 36-59 mo | 5.6 [4.2 to 7.6] |
  H1N1 Flu A/Brisbane/59/2007 IVR-148, Post 36-59 mo | 320.0 [142.8 to 716.9] |
  H3N2 Flu A/Uruguay/716/2007/ X175-C, Post 36-59 mo | 780.2 [274.5 to 2217.2] |
  B Flu B/Florida/04/2006, Post 36-59 mo | 59.4 [13.5 to 262.5] |

4. Other Pre Specified Outcome: Percentage of Participants With Influenza Titers ≥ 1:40 After Fluzone® Vaccination (Seroprotection)
Description: Seroprotection was defined as a post-vaccination Hemagglutination inhibition titer ≥ 1:40. Data presented for all participants and those enrolled at age 6 to 35 months.
Time Frame: Day 28 post-single dose or Day 21 post-Dose 2
Population: Seroprotection post-vaccination were determined in the per-protocol population.
  One each of the enrolled participants in the Primed and Naive groups, respectively, did not have valid post-vaccination serology test data.
Measure: Number; unit: Percentage of participants
Arm/Group | Primed Group | Naive/Inadequately Primed Group
Number analyzed (Participants) | 23 | 7
Percentage of participants
  H1N1 Flu A/Brisbane/59/2007 IVR-148 - All | 100 | 100
  H3N2 Flu A/Uruguay/716/2007/X175-C - All | 100 | 86
  B Flu B/Florida/04/2006 - All | 44 | 71
  H1N1 Flu A/Brisbane/59/2007 IVR-148 - 6-35 mo | 100 | 100
  H3N2 Flu A/Uruguay/716/2007/X175-C - 6-35 mo | 100 | 86
  B Flu B/Florida/04/2006 - 6-35 mo | 31 | 71

5. Primary Outcome: Number of Participants With Solicited Local and Systemic Reactions After Fluzone® Vaccination 2
Description: as for outcome 1
Time Frame: Day 0 to Day 3 post-vaccination 2
Population: Safety analysis (post-vaccination 2) was on all enrolled and vaccinated participants with available data, intent-to-treat population. (Data is part of Primary Outcome 1, no data were generated for the Primed Group)
Measure: Number; unit: Participants
Arm/Group | Primed Group | Naive/Inadequately Primed Group
Number analyzed (Participants) | 0 | 8
Participants
  Any Solicited injection site reaction |  | 3
  Any Tenderness |  | 1
  Grade 3 Tenderness (Cries when limb is moved) |  | 0
  Any Pain |  | 2
  Grade 3 Pain (Incapacitating) |  | 0
  Any Erythema |  | 1
  Grade 3 Erythema (≥ 5cm) |  | 0
  Any Swelling |  | 2
  Grade 3 Swelling (≥ 5cm) |  | 0
  Any Solicited Systemic Reaction |  | 4
  Any Fever |  | 2
  Grade 3 Fever (> 103.1 ºF) |  | 0
  Any Vomiting |  | 0
  Grade 3 Vomiting (≥ 6 Episode per 24 hour) |  | 0
  Any Crying Abnormal |  | 2
  Grade 3 Crying Abnormal (> 3 hours) |  | 0
  Any Drowsiness |  | 1
  Grade 3 Drowsiness (Sleeps most of the time) |  | 0
  Any Appetite Lost |  | 0
  Grade 3 Appetite Lost (Refuses ≥ 3 meals/feeds) |  | 0
  Any Irritability |  | 1
  Grade 3 Irritability (Inconsolable) |  | 0
  Any Headache |  | 0
  Grade 3 Headache (Prevents daily activities) |  | 0
  Any Malaise |  | 1
  Grade 3 Malaise (Prevents daily activities) |  | 0
  Any Myalgia |  | 1
  Grade 3 Myalgia (Prevents daily activities) |  | 0

6. Other Pre Specified Outcome: Percentage of Participants With Influenza Titers ≥ 1:40 After Fluzone® Vaccination (Seroprotection)
Description: Seroprotection was defined as a post-vaccination Hemagglutination inhibition titer ≥ 1:40. Data presented for participants enrolled at age 36 to 59 months.
Time Frame: Day 28 post-single dose or Day 21 post-Dose 2
Population: Seroprotection post-vaccination were determined in the per-protocol population. (Data is part of Outcome 5, no data were generated for the Naive/Inadequately Primed Group).
  One of the enrolled participants in the Primed groups did not have valid post-vaccination serology test data.
Measure: Number; unit: Percentage of participants
Arm/Group | Primed Group | Naive/Inadequately Primed Group
Number analyzed (Participants) | 23 | 0
Percentage of participants
  H1N1 Flu A/Brisbane/59/2007 IVR-148, 36-59 mo | 100 |
  H3N2 Flu A/Uruguay/716/2007/ X175-C, 36-59 mo | 100 |
  B Flu B/Florida/04/2006, 36-59 mo | 71 |

7. Other Pre Specified Outcome: Percentage of Participants With at Least a 4-Fold Rise in Influenza Titers After Fluzone® Vaccination (Seroconversion)
Description: Seroconversion was defined as a ≥ 4-fold increase in post-vaccination Hemagglutination inhibition titer. Data presented for all participants and those enrolled at age 6 to 35 months of age.
Time Frame: Day 28 post-single dose or Day 21 post-Dose 2
Population: Four-fold rises in vaccine Influenza titers were determined in the per-protocol population.
  One each of the enrolled participants in the Primed and Naive groups, respectively, did not have valid post-vaccination serology test data.
Measure: Number; unit: Percentage of participants
Arm/Group | Primed Group | Naive/Inadequately Primed Group
Number analyzed (Participants) | 23 | 7
Percentage of participants
  H1N1 Flu A/Brisbane/59/2007 IVR-148 - All | 50 | 86
  H3N2 Flu A/Uruguay/716/2007/X175-C - All | 91 | 86
  B Flu B/Florida/04/2006 - All | 41 | 71
  H1N1 Flu A/Brisbane/59/2007 IVR-148 - 6-35 mo | 50 | 86
  H3N2 Flu A/Uruguay/716/2007/X175-C - 6-35 mo | 94 | 86
  B Flu B/Florida/04/2006 - 6-35 mo | 31 | 71

8. Other Pre Specified Outcome: Percentage of Participants With at Least a 4-Fold Rise in Influenza Titers After Fluzone® Vaccination (Seroconversion)
Description: Seroconversion was defined as a ≥ 4-fold increase in post-vaccination Hemagglutination inhibition titer. Data presented for participants enrolled at age 36 to 59 months.
Time Frame: Day 28 post-single dose or Day 21 post-Dose 2
Population: Fold-rises in vaccine Influenza titers were determined in the per-protocol population. (Data is part of Outcome 7, no data were generated for the Naive/Inadequately Primed Group).
  One of the enrolled participants in the Primed groups did not have valid post-vaccination serology test data.
Measure: Number; unit: Percentage of participants
Arm/Group | Primed Group | Naive/Inadequately Primed Group
Number analyzed (Participants) | 23 | 0
Percentage of participants
  H1N1 Flu A/Brisbane/59/2007 IVR-148, 36-59 mo | 50 |
  H3N2 Flu A/Uruguay/716/2007/X-175-C, 36-59 mo | 83 |
  B Flu B/Florida/04/2006, 36-59 mo | 67 |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through the entire study, 1 or 2 months
Arm/Group | Primed Group | Naive/Inadequately Primed Group
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/8
Other Adverse Events (participants affected / at risk) | 4/24 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primed Group (N=24) | Naive/Inadequately Primed Group (N=8)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications